CLINICAL TRIAL: NCT01870076
Title: Effectiveness of Healing Touch on Sleep, Pain, Anxiety, Anesthesia Emergence, Satisfaction and Cost of Care in Surgical
Brief Title: The Effect of Healing Touch on Sleep
Acronym: Sleep7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Research Scientist, Shriners Hospitals for Children
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-1253
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Elective Reconstructive Surgery Population
MeSH Terms: interventions — Touch; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healing Touch Intervention (Experimental): Healing Touch performed one hour prior to bed.
  Interventions: Behavioral: Healing Touch
- Healing Touch Sham (Sham Comparator): Healing Touch Sham provided one hour prior to bed.
  Interventions: Behavioral: Healing Touch, Sham
- Control, Presence (Active Comparator): Control, Presence Intervention in the room one hour prior to bed.
  Interventions: Behavioral: Control, Presence
- Control, No Presence (No Intervention): No Presence in the room one hour prior to bed.

INTERVENTIONS:
Behavioral: Healing Touch
  Arms: Healing Touch Intervention
Behavioral: Healing Touch, Sham
  Arms: Healing Touch Sham
Behavioral: Control, Presence
  Arms: Control, Presence

SUMMARY:
Healing Touch improves measures of sleep the night prior to surgery, thus improving surgery-related morbidity.

DETAILED DESCRIPTION:
Patients are to randomized into one of 4 treatment groups upon enrollment. Depending on randomization group, the study participant receives the treatment the evening before elective surgery. A polysomnographic sleep study is then completed. Plan is to review the effect of the treatment group on sleep quantity and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. 5-25 years of age, inclusive
2. Elective admission for a reconstructive operative procedure
3. Planned use of general anesthesia during the elective operative procedure
4. Written informed consent, assent and Health Insurance Portability and Accountability Act (HIPAA) release signed by parent or legal guardian

Exclusion Criteria:

1. History of anoxic or suspected brain injury
2. History of head injury within the last year
3. Pre-existing neurological disorder
4. History of Reynaud's syndrome
5. Intellectual disability or inability to follow directions
6. Face/head phenomena that prevent(s) proper placement of polysomnography(PSG) leads
7. Taking medication for diagnosis of cardiomyopathy

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Gottschlich, PhD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The elective surgery patient list was assess for eligible patients. Those scheduled patient meeting inclusion criteria between 5-25 years of age were invited to participate in the study.
Pre-assignment Details: Upon verbal agreement, study randomization was assigned and a study consent was mailed to the patient. Arrangements for arrival time the night before surgery for the study procedures were made. After arrival to the unit the guardian reviewed the consent with study staff and upon written consent, study procedures began based on randomization.
Groups:
- Healing Touch Intervention: Healing Touch performed one hour prior to bed.
  Healing Touch
- Healing Touch Sham: Healing Touch Sham provided one hour prior to bed.
  Healing Touch, Sham
- Control, Presence: Control, Presence Intervention in the room one hour prior to bed.
  Control, Presence
Period: Overall Study
Arm/Group | Healing Touch Intervention | Healing Touch Sham | Control, Presence | Control, No Presence
Started | 10 | 12 | 8 | 11
Completed | 9 | 12 | 7 | 11
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healing Touch Intervention | Healing Touch Sham | Control, Presence | Control, No Presence | Total
Number analyzed (Participants) | 10 | 12 | 8 | 11 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 12 | 6 | 8 | 35
  Between 18 and 65 years | 1 | 0 | 2 | 3 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 4 | 23
  Male | 4 | 5 | 2 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 2 | 7
  White | 5 | 9 | 4 | 7 | 25
  More than one race | 1 | 3 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Number of Participants with Acuity Level 1 [Count of Participants; unit: Participants] — Level 1 is defined as same day surgery and observation (e.g. patients are technically never admitted as inpatient).
  Participants | 3 | 7 | 5 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Healing Touch Will Improve Total Sleep Time
Description: Data from nocturnal polysomnography, specifically total number of minutes of sleep time, will be compared between the healing touch and non healing touch groups.
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Healing Touch Intervention | Healing Touch Sham | Control, Presence | Control, No Presence
Number analyzed (Participants) | 9 | 12 | 7 | 11
minutes | 352.9 (17.0) | 368.2 (22.8) | 383.1 (26.4) | 367.2 (19.3)

2. Secondary Outcome: Preoperative Cortisol Level
Description: Cortisol level was compared among the 4 study groups.
Time Frame: Labs were drawn immediately pre-op.
Population: Surgical patients who completed Polysomnography and pre-op study labs.
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Healing Touch Intervention | Healing Touch Sham | Control, Presence | Control, No Presence
Number analyzed (Participants) | 9 | 12 | 7 | 11
mcg/dL | 6.7 (4.2) | 7.1 (4.3) | 6.9 (3.4) | 17.7 (34.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Healing Touch Intervention | Healing Touch Sham | Control, Presence | Control, No Presence
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT01870076/Prot_SAP_000.pdf